CLINICAL TRIAL: NCT05017194
Title: Efficacy and Safety of Emodepside in Adults Infected With Trichuris Trichiura and Hookworm: Randomized Two Stages Phase II Seamless Adaptive Controlled Single-blind Trials
Brief Title: Efficacy and Safety of Emodepside in Adults Infected With Trichuris Trichiura and Hookworm
Acronym: EMODEP_PEMBA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jennifer Keiser (Other)
Collaborators: Public Health Laboratory Ivo de Carneri (Other)
Responsible Party: Sponsor-Investigator, Jennifer Keiser, Prof. Dr., Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMODEP_PEMBA
Record Dates: First submitted 2021-07-05; First posted 2021-08-23 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Trichuris Trichiura; Infection; Hookworm Infections
Keywords: Emodepside; Trichuris trichiura; Hookworm; Soil-transmitted helminths; Efficacy; Safety; Dose selection
MeSH Terms: conditions — Trichuriasis; Hookworm Infections; Ancylostomiasis | interventions — emodepside

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Emodepside 5 mg (Experimental)
  Interventions: Drug: Emodepside
- Emodepside 10 mg (Experimental)
  Interventions: Drug: Emodepside
- Emodepside 15 mg (Experimental)
  Interventions: Drug: Emodepside
- Emodepside 20 mg (Experimental)
  Interventions: Drug: Emodepside
- Emodepside 25 mg (Experimental)
  Interventions: Drug: Emodepside
- Emodepside 30 mg (Experimental)
  Interventions: Drug: Emodepside
- Albendazole (Active Comparator)
  Interventions: Drug: Emodepside
- Placebo (Placebo Comparator)
  Interventions: Drug: Emodepside

INTERVENTIONS:
Drug: Emodepside — Treatment with ascending doses of emodepside (from 5 mg to 30 mg) or albendazole (400 mg) or placebo.

SUMMARY:
The rationale of the study is to provide evidence on the efficacy and safety of Emodepside in adults infected with Trichuris trichiura and hookworm.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged between 18 and 45 years
* Written and signed informed consent
* Examined by a study physician before treatment
* Provided two stool samples at baseline
* Trichuris trichiura and hookworm EPG ≥ 48 and at least two Kato-Katz thick smears slides with more than one Trichuris trichiura and hookworm eggs

Exclusion Criteria:

* Pregnant or lactating and/or planning to become pregnant within three months after drug treatment
* Type 1 and/or 2 diabetes
* Psychiatric disorders
* History of ophthalmological conditions
* Presence or history of major systemic or chronic illnesses, as assessed by a medical doctor, during initial clinical assessment
* Suffers from severe anaemia (Hb < 80 g/l)
* Received anthelminthic treatment within past four weeks
* Attending other clinical trials during the study
* Received strong CYP3A4 inducers or inhibitors as well as concomitant treatments that are relevant substrate for CYP3A4 such as clarithromycin, erythromycin and rifampicin
* Received strong P-gp inhibitors as well as concomitant treatments that are relevant substrates for P-gp such as clotrimazole and ritonavir

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 442 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Cure rate (CR) of emodepside against Trichuris trichiura | In the week between 14 and 21 days post-treatment
  CR will be calculated as the percentage of Trichuris trichiura egg-positive participants at baseline who become egg-negative after treatment.
Cure rate (CR) of emodepside against hookworm | In the week between 14 and 21 days post-treatment
  CR will be calculated as the percentage of hookworm egg-positive participants at baseline who become egg-negative after treatment.

SECONDARY OUTCOMES:
Geometric Mean Egg Reduction Rate (ERR) of the emodepside against Trichuris trichiura and hookworm. | In the week between 14 and 21 days post-treatment
  Eggs per gram of stool (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. The egg reduction rate (ERR) is calculated as follows: ERR = (1-(geometric mean EPG at follow-up/geometric mean EPG at baseline))*100). Note: in contrast to the publication the "outcome measure" entry mask requires the complementary percentage: (geometric mean at follow-up/geometric mean at baseline)*100).
CR against Ascaris lumbricoides | In the week between 14 and 21 days post-treatment
  CR will be calculated as the percentage of Ascaris lumbricoides egg-positive participants at baseline who become egg-negative after treatment.
ERR against Ascaris lumbricoides | In the week between 14 and 21 days post-treatment
  Eggs per gram of stool (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. The egg reduction rate (ERR) is calculated as follows: ERR = (1-(geometric mean EPG at follow-up/geometric mean EPG at baseline))*100). Note: in contrast to the publication the "outcome measure" entry mask requires the complementary percentage: (geometric mean at follow-up/geometric mean at baseline)*100).

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Laboratory - Ivo de Carneri, Chake Chake, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Montresor A, Gabrielli AF. Emodepside - A Promising Drug for the Treatment of Soil-Transmitted Helminthiases. N Engl J Med. 2023 May 18;388(20):1907-1908. doi: 10.1056/NEJMe2303793. No abstract available. PMID 37195949
- [Derived] Mrimi EC, Welsche S, Ali SM, Hattendorf J, Keiser J. Emodepside for Trichuris trichiura and Hookworm Infection. N Engl J Med. 2023 May 18;388(20):1863-1875. doi: 10.1056/NEJMoa2212825. PMID 37195942